CLINICAL TRIAL: NCT03463928
Title: Phase I Study to Evaluate Treatment of Relapsed or Refractory Leukemia With Donor-derived HSCT Following Donor-derived CD19/22 Bispecific CAR-T Cells or CD19-directed CAR-T Cells
Brief Title: A Feasibility and Safety Study of Concomitant Therapy With Allo-CAR-T Cells and Allo-HSCT in Patients With Relapse or Refractory Leukemia
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Han weidong, Director of Molecular & Immunological Department, Biotherapeutic Department, Chinese PLA General Hospital, Chinese PLA General Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHN-PLAGH-BT-027
Record Dates: First submitted 2018-03-07; First posted 2018-03-13 (Actual); Last update posted 2018-03-13 (Actual); Status verified 2018-03

CONDITIONS: B Cell Leukemia
MeSH Terms: conditions — Leukemia, B-Cell

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: donor-derived CD19/22 bispecific CAR-T cells or CD19-directed CAR-T cells; donor-derived-HSCT — The allo-CAR-T cells will be infused in a fractionated manner, 1/3 on day 0, 2/3 on day 1.The allo-HSCT will be infused on day 2.

SUMMARY:
Allogenic hematopoietic stem cell transplant (Allo-HSCT) is routinely used for treatment of aggressive hematological malignancies. The biological foundation of allo-HSCT is the graft-versus-leukemia (GVL) effect, which is primarily mediated by donor T cells present in the graft and is able to eradicate malignant B cells either CD19+ or CD19-. Relapse following an allo-HSCT remains a major challenge in the treatment of B-ALL. CD19-directed CAR-T cell therapy has shown promising results for the treatment of relapsed or refractory B-cell malignancies; however, a subset of patients relapse due to the loss of CD19 in tumor cells. Co-infusion of donor-derived CD19/22 bispecific CAR-T cells or CD19-directed CAR-T cells and donor-derived-HSCT has the potential to combine the CAR-T cell mediated targeted elimination of CD19 expressing B cells with GVL effect, which could have clear advantages in reducing the risk of relapse and the evolution of CD19- escape variants or clonally related malignancies in other lineages. Therefore, a complete and durable tumor responses induced by this immunotherapy could be expected.

DETAILED DESCRIPTION:
1. PRIMARY OBJECTIVES:

   1. To evaluate the feasibility and safety of donor-derived HSCT following donor-derived CD19/22 bispecific CAR-T cells or CD19-directed CAR-T cells in patients with relapsed or refractory leukemia.
   2. To evaluate the duration of in vivo persistence of adoptively transferred CAR-T cells, and the phenotype of persisting T cells. Real Time polymerase chain receptor (RT-PCR) and Flow cytometry(FCM) analysis of PB,BM will be used to detect and quantify survival of infused allo-CAR-T cells over time.
   3. To evaluate the donor chimerism after co-infusion of donor-derived CD19/22 bispecific CAR-T cells or CD19-directed CAR-T cells and donor-derived-HSCT
2. SECONDARY OBJECTIVES:

   1. For patients with detectable disease, measure anti-tumor response due to co-infusion of donor-derived CD19/22 bispecific CAR-T cells or CD19-directed CAR-T cells and donor-derived-HSCT.

The allo-CAR-T cells will be infused in a fractionated manner, 1/3 on day 0, 2/3 on day 1.The allo-HSCT will be infused on day 2.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participant
2. 12 Years to 60 Years
3. Patient with relapsed or refractory B-cell leukemia or lymphoma
4. Estimated life expectancy ≥ 12 weeks (according to investigator's judgement)
5. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1
6. Adequate organ function

Exclusion Criteria:

1. Prior malignancy, except carcinoma in situ of the skin or cervix treated with curative intent and with no evidence of active disease
2. Diagnosis of Burkitt's leukemia/lymphoma according to WHO classification or chronic myelogenous leukemia lymphoid blast crisis
3. Richter's syndrome
4. Presence of Grade II-IV (Glucksberg) or B-D (IBMTR) acute or extensive chronic GVHD at the time of screening
5. Subjects with any autoimmune disease or any immune deficiency disease or other disease in need of immunosuppressive therapy
6. Severe active infection (uncomplicated urinary tract infections, bacterial pharyngitis is allowed), Prophylactic antibiotic, antiviral and antifungal treatment is permissible
7. Active hepatitis B, active hepatitis C, or any human immunodeficiency virus (HIV) infection at the time of screening
8. Patient has an investigational medicinal product within the last 30 days prior to screening
9. Previous treatment with investigational gene or cell therapy medicine products
10. Concurrent use of systemic steroids. Recent or current use of inhaled steroids is not exclusionary
11. Pregnant or nursing women

Ages: 12 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Estimated)
Dates: Start 2017-10-08 (Actual); Primary Completion 2019-06 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Severe/Adverse Events as a Measure of Safety and Tolerability | 24 weeks

SECONDARY OUTCOMES:
Overall remission rate (ORR) = CR + CRi | 24 weeks
Six-month Overall survival | 24 weeks
Six-month Progression free survival | 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Biotherapeutic Department and Hematology Department of Chinese PLA General Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No